CLINICAL TRIAL: NCT00963963
Title: Reducing HIV Risks in African American Teens in High Poverty Urban Settings
Brief Title: Reducing HIV Risks in African American Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education Development Center, Inc. (Industry)
Responsible Party: Principal Investigator, Lydia O'Donnell, Senior Scientist, Education Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD054297 (NIH)
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: HIV Infections
Keywords: sexual health; adolescent health; parent education; HIV Seronegativity; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- health promotion materials (Active Comparator): Parents receive health promotion booklets
  Interventions: Behavioral: Healthy Futures parent education
- attention-controlled parent print materials (Active Comparator): Booklets on adolescent sexuality and health
  Interventions: Behavioral: Healthy Futures parent education
- audio-CD parent education (Experimental): audio-CDs on parenting practices
  Interventions: Behavioral: Healthy Futures parent education

INTERVENTIONS:
Behavioral: Healthy Futures parent education — Multi-year audio CD parent education

SUMMARY:
This study is developing and testing an innovative, parent education intervention, Preparing Our Sons and Daughters for Healthy Futures. This intervention aims to reduce HIV risk among African American and other Black youth living in high-poverty urban neighborhoods. Investigators, working with a community advisory board and focus groups of youth and parents, will develop a multi-year set of audio-CDs to promote positive parenting practices that support young adolescents in establishing healthy patterns of behavior. This parent education intervention will be tested in a field trial with families of 6th graders recruited from multiple schools in New York City. Baseline and annual follow up surveys will be conducted until youth enter high school. Families receiving the intervention will be compared to those assigned to either an attention-controlled print materials condition or a non-attention controlled condition. It is hypothesized that youth whose parents receive the intervention will delay sexual initiation and report fewer sexual risks, and that their parents will report more positive parenting practices.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at selected schools
* 6th graders and their parents

Exclusion Criteria:

* Non-English speaking

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2013-04-30 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
youth risk behaviors | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Education Development Center, Newton, Massachusetts, United States